CLINICAL TRIAL: NCT00874354
Title: REVITALIZE: Randomized Evaluation of Intracoronary Transplantation of Bone Marrow Stem Cells in Myocardial Infarction
Brief Title: Randomized Evaluation of Intracoronary Transplantation of Bone Marrow Stem Cells in Myocardial Infarction
Acronym: REVITALIZE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Raj Makkar, Director, Interventional Cardiology and Cardiac Catheterization Laboratory, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4441
Record Dates: First submitted 2007-12-26; First posted 2009-04-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Heart Attack; Infarct; Stem Cells; Bone Marrow Derived Mononuclear Cells; CHF; Congestive Heart Failure; Stent; PCI; Percutaneous Coronary Intervention
MeSH Terms: conditions — Myocardial Infarction; Infarction; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous bone marrow stem cells (Experimental): Patients within 3 to 14 days from percutaneous coronary intervention (PCI) and stent implantation for Acute Myocardial Infarction (AMI) will receive either 50 cc's or 100 cc's of autologous bone marrow mononuclear cells through an intracoronary tranplantation of stem cells into the infarct-related coronary artery.
  Interventions: Drug: Intracoronary Transplantation of Bone Marrow Stem Cells

INTERVENTIONS:
Drug: Intracoronary Transplantation of Bone Marrow Stem Cells — Intracoronary application of autologous bone marrow-derived mononuclear cells in infarct artery 3 - 14 days after PCI for acute myocardial infarction.
  Other Names: REVITALIZE

SUMMARY:
This research is being done because currently there is no effective way in regenerating or replacing the heart muscle that has been damaged after a heart attack.

The purpose of this study is to test whether injecting cells obtained from the patient's bone marrow into the coronary artery can regenerate and replace heart tissue to strengthen heart and prevent heart from dilating and developing heart failure.

DETAILED DESCRIPTION:
The main objective of this study is to investigate the safety and clinical outcome of intracoronary infusion of autologous bone marrow cells in patients with myocardial infarction (MI). We hypothesize that patients treated with stem cell therapy will have beneficial effects on left ventricular (LV) remodeling and functional regeneration after MI and successful primary percutaneous coronary intervention (PCI) in setting of prospective randomized controlled trial.

Congestive heart failure (CHF), which is most commonly caused by acute myocardial infarction (AMI), is the most frequent cause of hospitalization in the United States in patients over the age of 65. Although current pharmacotherapy can inhibit neurohormonal activation, this falls short in preventing LV remodeling and the development of CHF. Stem cells are undifferentiated pluripotent cells that can be obtained from the patient and have the potential to proliferate and differentiation into cardiomyocytes. The majority of the data on stem cell transplantation comes from preclinical animal studies. Although the results are interesting and perhaps safe, early phase I clinical studies are small and are very preliminary. Data from large, randomized controlled trials are needed to clarify the short and long term effects of cellular cardiomyoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myocardial infarction (ST elevation in at least 2 leads ≥ 0.2 mV in V1,V2 or V3 or ≥ 0.1 mV in other leads), treated by one of the following procedures:

  * Acute PCI with stent implantation for acute ST elevation MI for either denovo lesions or in-stent thrombosis
  * Treatment with thrombolysis followed by PCI with stent implantation.
* Acute PCI / stent implantation has been successful (residual stenosis visually < 30% and TIMI flow ≥ 2).
* At the time of inclusion (≥ 1 day post PCI) patient does no longer require i.v. catecholamines or mechanical hemodynamic support (aortic balloon pump)
* Significant regional wall motion abnormality on echocardiography at the time of acute PCI (ejection fraction ≤ 50% on visual estimation).
* Maximal cardiac troponin elevation ≥ 4 (measured at 37° C)
* Age 18 - 80 Years
* Written informed consent

Exclusion Criteria:

* Regional wall motion abnormality outside the area involved in the index acute myocardial infarction.
* Need to acutely revascularize additional vessels, outside the infarct artery.
* Arteriovenous malformations or aneurysms
* Active infection or fever or diarrhea within last 4 weeks.
* Chronic inflammatory disease
* HIV infection or active hepatitis
* Neoplastic disease without documented remission within the past 5 years.
* Cerebrovascular insult within 3 months
* Impaired renal function (creatinine > 2 mg/dl) at the time of cell therapy
* Significant liver disease (GOT > 2x upper limit) or spontaneous INR > 1.5)
* Anemia (hemoglobin < 8.5 g/dl)
* Platelet count < 100,000/µl
* Hypersplenism
* History of bleeding disorder
* Gastrointestinal bleeding within 3 months
* Major surgical procedure or trauma within 2 months
* Uncontrolled hypertension
* Pregnancy
* Mental retardation
* Previously performed stem / mononuclear cell therapy
* Participation in another clinical trial within the last 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of intracoronary administration of autologous bone marrow-derived mononuclear cells; Improvement of global left ventricular ejection fraction by cardiac MRI and echocardiography after 4 months. | 4 months from procedure

SECONDARY OUTCOMES:
Freedom from Major Adverse Cardiac Event (MACE) | 12 months from procedure

CONTACTS AND LOCATIONS:
Overall Officials: Raj Makkar, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No